CLINICAL TRIAL: NCT04082559
Title: Biomarker-based Multidisciplinary Team Approach to Personalized Microbial-targeted Treatment of Pouchitis and Crohn's Disease
Brief Title: Biomarker-based Multidisciplinary Team (Bio-MDT) Approach to Personalized Microbial-targeted Treatment of Pouchitis and Crohn's Disease
Acronym: Bio-MDT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Tel Aviv University (Other)
Responsible Party: Principal Investigator, IRIS DOTAN, Head of The Gastroenterology Division, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0129-19-RMC
Record Dates: First submitted 2019-08-28; First posted 2019-09-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Ciprofloxacin; Metronidazole; Doxycycline; Anti-Bacterial Agents; Diet; WW Domain-Containing Oxidoreductase; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antibiotic treatment (Other): Patients with active disease will be randomized and will receive a prescription for one of two antibiotic regimens.
  1. Ciprofloxacin 500 mg 2/d + metronidazole 500 mg 2/d for two weeks
  2. Doxycycline 100 mg 2/d + metronidazole 500 mg 2/d for two weeks
  Interventions: Other: Arm 1- Antibiotics treatment; Other: Arm 2- Antibiotics treatment
- Combination therapy (Antibiotics + diet) (Other): 1. Favorable antibiotics (according to aim 1) for two weeks + Mediterranean diet (MED) for 8 weeks.
  2. Favorable antibiotics (according to aim 1) for two weeks + specific carbohydrate diet (SCD) for 8 weeks.
  Interventions: Other: Arm 1- Combination therapy (Antibiotics + diet); Other: Arm 2- Combination therapy (Antibiotics + diet)
- Nutritional prevention (Other): Patients in clinical remission will be recruited to a dietary prevention study.
  1. Mediterranean diet
  2. Control- based on the American Dietetic Association recommendations for patients with IBD
  3. Personalized nutrition group- based on prior results from study- NCT02858557
  Interventions: Other: Arm 1- Nutritional prevention; Other: Arm 2- Nutritional prevention; Other: Arm 3- Nutritional prevention

INTERVENTIONS:
Other: Arm 1- Antibiotics treatment — Patients with active disease will be randomized and will receive a prescription antibiotic regimens
  Other Names: Ciprofloxacin 500 mg 2/d + metronidazole 500 mg 2/d for two weeks
  Arms: Antibiotic treatment
Other: Arm 2- Antibiotics treatment — Patients with active disease will be randomized and will receive a prescription antibiotic regimens
  Other Names: Doxycycline 100 mg 2/d + metronidazole 500 mg 2/d for two weeks
  Arms: Antibiotic treatment
Other: Arm 1- Combination therapy (Antibiotics + diet) — Patients with active disease receiving a prescription for the antibiotic regimen defined as favorable in the antibiotics according to aim 1 , and randomized into one of two dietary interventions: Mediterranean diet (MED) or the specific carbohydrate diet (SCD).
  Other Names: Favorable antibiotics (according to aim 1) for two weeks + Mediterranean diet (MED) for 8 weeks.
  Arms: Combination therapy (Antibiotics + diet)
Other: Arm 2- Combination therapy (Antibiotics + diet) — Patients with active disease receiving a prescription for the antibiotic regimen defined as favorable in the antibiotics according to aim 1 , and randomized into one of two dietary interventions: Mediterranean diet (MED) or the specific carbohydrate diet (SCD).
  Other Names: Favorable antibiotics (according to aim 1) for two weeks + specific carbohydrate diet (SCD) for 8 weeks.
  Arms: Combination therapy (Antibiotics + diet)
Other: Arm 1- Nutritional prevention — Patients in clinical remission will be recruited to a dietary prevention study
  Other Names: Mediterranean diet
  Arms: Nutritional prevention
Other: Arm 2- Nutritional prevention — Patients in clinical remission will be recruited to a dietary prevention study
  Other Names: Control- based on the American Dietetic Association recommendations for patients with IBD
  Arms: Nutritional prevention
Other: Arm 3- Nutritional prevention — Patients in clinical remission will be recruited to a dietary prevention study
  Other Names: Personalized nutrition group- based on prior results from study- NCT02858557
  Arms: Nutritional prevention

SUMMARY:
Crohn's disease (CD) and ulcerative colitis (UC) are chronic inflammatory bowel diseases (IBD) currently affecting over 5 million patients globally, mostly young adults. These conditions are often debilitating, disabling and may markedly affect patient's quality of life. Despite important advances in research, the pathogenesis of IBD remains obscure, the incidence-rising, the condition - incurable, and drugs have a modest effect. The common denominator may be environmental factors, specifically diet and the microbiome, which remain a fundamental unmet need in IBD care as high quality randomized trials and mechanistic research are limited. Up to a quarter of patients with UC may undergo complete large bowel resection due to disease complications. In order to preserve bowel continuity, this surgery includes a restorative part with creation of a reservoir ("pouch") from normal small bowel instead of the resected rectum. The majority of these patients develop small intestinal inflammation in the previously normal small bowel creating the pouch ("pouchitis").

Based on our results from previous studies, we hypothesized that personalized antibiotics and dietary interventions will modify microbial composition and result in significantly improved outcomes, specifically resolution of inflammation and prolonged remission rates in patients with a pouch.

Aims:

1. Compare the effect of two antibiotic treatments on clinical, inflammatory and microbiological outcomes of patients with pouch inflammation.
2. Evaluate the effect of combined microbiome-targeted antibiotic and dietary intervention as treatment and prevention strategy in patients after pouch surgery.
3. Evaluate the effect of a microbiome-targeted dietary intervention as prevention strategy in patients after pouch surgery.
4. Identify predictors for response to specific antibiotic and dietary interventions.

DETAILED DESCRIPTION:
All patients will undergo comprehensive screening by the bio-MDT.

Aim 1: Antibiotic treatment- (patients with active disease) will be randomized to receive a prescription for one of two antibiotic regimens.

1. Ciprofloxacin + metronidazole
2. Doxycycline+ metronidazole

Aim 2: Combination therapy ( Antibiotics+diet) After arm 1 recruitment completion, a favorable antibiotic regimen will be determined and recommended in arm 2, in which, patients with active disease will be randomized to

1. Favorable antibiotics + Mediterranean diet (MED)
2. Favorable antibiotics + The Specific Carbohydrate Diet (SCD)

Aim 3: Nutritional prevention-

Patients in clinical remission will be recruited to a dietary prevention study and be allocated to one of three groups:

1. Mediterranean diet (MED)
2. Control- based on the American Dietetic Association recommendations for patients with IBD.
3. Personalized nutrition group- based on prior results from study- NCT02858557

Comprehensive assessment including nutritional, clinical, inflammatory and microbial parameters will be performed at baseline and at weeks 2,3,4,8,26, 52.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are able and willing to sign an informed consent
2. Patients with UC who underwent pouch surgery and have a functioning pouch
3. Disease activity (PDAI and PGA) according to study arm 1-3 inclusion

Exclusion Criteria:

1. Patients with ileostomy
2. Significant comorbidity that precludes the patient from participating according to the physicians' judgment
3. Non-Hebrew readers
4. Pregnant and lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-06-11 (Estimated); Study Completion 2023-06-11 (Estimated)

PRIMARY OUTCOMES:
Time interval to response | One year
  Decrease in PGA and PDAI
Time interval to remission | One year
  PGA=0 and PDAI<7

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided